CLINICAL TRIAL: NCT06734689
Title: Genetic Determinants of Myocarditis Induced by Immune-checkpoint Inhibitors
Acronym: GICICA-Control
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220921; 2024-A00410-47 (Other: ANSM)
Record Dates: First submitted 2024-11-05; First posted 2024-12-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: ICI-myocarditis
Keywords: Myocarditis; Myositis; Immune-checkpoint inhibitors; Pharmacogenetic
MeSH Terms: conditions — Myocarditis; Myositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ICI-tolerant patients without suspicion of myotoxicity (Controls): 300 Patients on ICI since at least 3 months with a minimum of 2 ICI doses received having no appearance (as compared to baseline known pre-ICI) of new cardio-muscular symptoms or ECG abnormality or wall motion abnormality or troponin-T increase (above Upper Limit of Normal if normal prior to ICI start, or over twice its troponin-T baseline value if abnormal before ICI start)
- Patients with refuted suspicion of ICI-myocarditis (controls): 100 Cancer patients treated with ICI and with definite ICI-induced myocarditis according to last updated diagnostic criteria's
- ICI-Myocarditis Cases (Cases): 100 Cancer patients treated with ICI admitted for a suspicion of ICI-myocarditis subsequently infirmed

SUMMARY:
Immune checkpoint inhibitors (ICI) are active in multiple cancers. Their main drawback is the incidence of immune related adverse events; among which ICI-myocarditis (ICIM) is rare but can be the most life-threatening (up to 50% lethal). ICIM is due to ICI unleashing cytotoxic auto-reactive T-cells recognizing a culprit target antigen located on muscles and destroying them. Most often, ICIM occurs within a systemic ICI-myotoxicity, with peripheral muscular involvement (ICI-myositis), mimicking eventually myasthenia-gravis syndrome. Human Leukocyte Antigen (HLA) are cell surface proteins key for the regulation of the immune system acting via presentation of culprit antigens by antigen presenting cells (macrophages) to T-cells, subsequently triggering the destruction/tolerance of cells carrying this antigen. The HLA system (chromosome 6) is the most polymorphic region in the human genome and is associated with auto-immunity including myocarditis. HLA class I alleles have been strongly associated with some T-cell-mediated drug hypersensitivity reactions with handful patients needed to be tested to prevent a single case, leading to globally required cost-effective HLA typing pre-prescription for some drugs.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICI) are revolutionary anticancer therapeutics indicated and active in multiple different cancer types. Approved ICI include antibodies targeting and blocking four main molecules, normally toning down immune system activation: CTLA4 (cytotoxic T-lymphocyte antigen 4), LAG3 (Lymphocyte Activation Gene-3), PD1 (Programmed cell Death protein 1) and its ligand (PDL1). Notably, a set of ~30-40 other molecules are considered as key in immune-checkpoint system and currently investigated as potential drug targets. A main drawback of ICI is the incidence of immune related adverse events (irAE), occurring after unleashing the immune system and which can potentially affect any organ and eventually be fatal. Among IrAE, myocarditis is rare (0.25-1% of ICI treated patients) but is the most life-threatening irAE (up to 50% mortality). ICI-myocarditis occur fast after ICI start (1-3 doses) and is mainly driven by T-cells and macrophages infiltrating muscles including the heart and leading to its necrosis, which manifest clinically with fatal arrhythmias and cardiogenic shock. Another key clinical feature of this myotoxic syndrome induced by ICI is the co-occurrence of ICI-myocarditis with ICI-myositis affecting virtually any other muscle (potentially mimicking ICI-myasthenia gravis), including the respiratory muscles which can lead to severe hypercapnia and death. This mechanism is triggered by ICI boosting a subset of cytotoxic T-cells recognizing a culprit muscular target antigen located on muscles. Co-occurrence of ICI-myocarditis with ICI-myositis has been reported to be almost universal (>90%) in a prospective consecutive cohort of 40 ICI-myocarditis with cardiac and muscular biopsies performed.

Human Leukocyte Antigen (HLA) are key cell-surface proteins responsible for the regulation of the immune system, notably by acting thru the presentation of culprit antigens by antigen presenting cells (e.g macrophages) to T-lymphocytes triggering the destruction/tolerance of cells carrying the culprit antigen in the organism. The HLA system (a complex of genes on chromosome 6) is the most polymorphic region/locus in the human genome and has been associated with protection and predisposition to a broad array of infectious, malignant, and autoimmune diseases including myocarditis. In the past two decades, HLA class I alleles have been strongly associated with T-cell-mediated drug hypersensitivity reactions. For example, in the case of abacavir hypersensitivity and HLA-B*57:01, the negative predictive value is 100% and there is low number of patients (dozens) needed to be tested to prevent a single case, which has led to a durable and effective global pre-prescription cost-effective screening strategy, required by regulatory such as FDA. Indeed, only 18 patients with abacavir associated hypersensitivity versus ~160 drug-tolerant were needed to identify the association with the HLA-B*57:01 allele that demonstrated a frequency of 78% in cases versus 2% in drug-tolerant controls. Similar examples with comparable magnitude of effects, i.e. high frequency (~30%-70%) of risk alleles in cases and low frequency (~2%) in controls, have been observed with various HLA (e.g., -B,-C,-A,-DRB1) alleles and auto-immune conditions (e.g., carbamazepine-Toxidermia, allopurinol-Toxidermia, flucloxacillin-hepatitis and statins-necrotizing myopathies).

Altogether, these observations have led us to hypothesize that the susceptibility to ICI-myocarditis could be under the influence of genetic factors within HLA genes but also elsewhere in the genome. Therefore, the investigators propose to perform a genetic study to identify common and rare variants associated with the risk of myocarditis induced by ICI in cancer patients.

The main hypothesis of this proposed work is that common and/or rare polymorphism with large effect size might predispose to the incidence of myocarditis/myotoxicities induced by immune-checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients on ICI since at least 3 months with a minimum of 2 ICI doses received having no appearance (as compared to baseline known pre-ICI) of a new cardio-muscular symptoms or ECG abnormality or WMA or troponin-T increase (above ULN if normal prior to ICI start, or over twice its troponin-T baseline value if abnormal before ICI start).
2. Signature of informed consent before any trial procedure from the patient
3. Patients covered by social security regimen (excepting AME).

Exclusion Criteria:

1. Age <18 years of age.
2. Pregnant or breast-feeding women
3. People under legal protection measure (safeguard measures)

Specific exclusion criteria for the magnetic resonance imaging sub-study (MRI)

* Patients with a contraindication to MRI (claustrophobia, some wearing equipment with magnetic properties: pacemaker, ferromagnetic equipment, etc.)
* Intolerance to gadolinium, or severe renal insufficiency (GFR<30 ml/min/1.73 m2).

Of note, the other groups of patients needed to complete this study; i.e the patients with refuted suspicion of ICI-myocarditis who will serve as controls, and the patients with ICI-myocarditis (cases) are included in another protocol (NCT05454527)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients treated by immune checkpoint inhibitors
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
Identify common and rare variants in HLA regions and elsewhere in the genome associated with ICI Myocarditis. | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  -Identify common single nucleotide variants(SNV) associated with ICI-myocarditis, such as variants in HLA regions with a genome-wide association study using 100 ICIM and 400 ICI-controls. Any association that reach the genome wide significance levels of 5.10-8 as well as any association mapping to candidate HLA and immune checkpoint genes with p-value<10-5 will be tested for replication in an external international validation cohort.
Identify common and rare variants in HLA regions and elsewhere in the genome associated with ICI | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  -Sequence the entire protein-coding regions of the genome of all patients to identify extremely rare SNV associated with a strong risk of ICI-myocarditis. Investigators will focus on the search of rare SNV that are present only in the group of ICI-myocarditis patients and prioritize those with high predicted deleteriousness and mapping to candidate genes (immunity genes,cardiac genes).Candidate variants/genes will be further explored in an international validation cohort and by functional studies using a mice model phenocopying ICI-myocarditis condition.

SECONDARY OUTCOMES:
Build a polygenic risk score (PRS) based on common variants to discriminate ICIM vs ICI-controls. | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  A PRS will be constructed using the combination of common polymorphisms associated with ICI-myocarditis
Study the impact of age, sex, type of cancer, type of immunotherapies, and race on the penetrance of identified risk-allele associated with ICI myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  A multivariable model integrating both the PRS together with clinical variable including age, sex, race, type of cancer, type of immunotherapies will be derived and its discriminatory capacities will be investigated using ROC (receiver operating characteristic) curves
Study the impact of age, sex, type of cancer, type of immunotherapies, and race on the penetrance of identified risk-allele associated with ICI myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  A multivariable model integrating both the PRS together with clinical variable including age, sex, race, type of cancer, type of immunotherapies will be derived and its discriminatory capacities will be investigated using NRI (Net reclassification index)
Study the impact of age, sex, type of cancer, type of immunotherapies, and race on the penetrance of identified risk-allele associated with ICI myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  A multivariable model integrating both the PRS together with clinical variable including age, sex, race, type of cancer, type of immunotherapies will be derived and its discriminatory capacities will be investigated using IDI (integrated discrimination improvement)
Calculation of the diagnostic properties of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  Compute the diagnostic properties (ROC curves) of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis by calculating number of patients to test to predict one ICI-myocarditis event
Calculation of the diagnostic properties of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  Compute the diagnostic properties (ROC curves) of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis by calculating sensitivity
Calculation of the diagnostic properties of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  Compute the diagnostic properties (ROC curves) of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis by calculating specificity
Calculation of the diagnostic properties of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  Compute the diagnostic properties (ROC curves) of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis by calculating positive predictive value
Calculation of the diagnostic properties of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  Compute the diagnostic properties (ROC curves) of any relevant SNV/PRS associated with ICI myocarditis vs. initially suspected and subsequently refuted ICI-myocarditis by calculating negative predictive value
Study the effects of ICI on peripheral muscles homeostasis in ICI-control | Peripheral muscle biopsies performed before ICI start and within 3 to 6 months after ICI start
  Study the histopathological changes (immune cells counts) in peripheral muscles of ICI control
Study the cardiac and diaphragmatic changes on ICI treatment | Examinations performed once before ICI start and within 3 to 6 months after ICI start
  Study the cardio muscular biomarkers circulating variations on ICI (troponin levels)
Study the cardiac and diaphragmatic changes on ICI treatment | Examinations performed once before ICI start and within 3 to 6 months after ICI start
  Study the cardio muscular biomarkers circulating variations on ICI (creatine-kinase levels)
Study the cardiac and diaphragmatic changes on ICI treatment | Examinations performed once before ICI start and within 3 to 6 months after ICI start
  Study the cardiac functional changes on ICI evaluated by echocardiography
Study the cardiac and diaphragmatic changes on ICI treatment | Examinations performed once before ICI start and within 3 to 6 months after ICI start
  Study the cardiac functional changes on ICI evaluated by magnetic resonance imaging
Study the cardiac and diaphragmatic changes on ICI treatment | Examinations performed once before ICI start and within 3 to 6 months after ICI start
  Study the diaphragmatic functional changes on ICI evaluated by echography
Study the cardiac and diaphragmatic changes on ICI treatment | Examinations performed once before ICI start and within 3 to 6 months after ICI start
  Study the diaphragmatic functional changes on ICI evaluated by magnetic resonance imaging
Construction of a PRS using the combination of common polymorphisms associated with ICI-cancer response | Baseline before ICI start and one follow-up point between 3 to 6 months after ICI
  A PRS will be constructed using the combination of common polymorphisms associated with ICI-cancer response

CONTACTS AND LOCATIONS:
Overall Officials: Joe Elie SALEM, Pr, Principal Investigator — Assitance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.